CLINICAL TRIAL: NCT05363917
Title: Phase II Double-Blinded, Placebo-Controlled Randomized Study Examining the Safety and Efficacy of Natrunix Versus Methotrexate (+Folate) for the Treatment of Rheumatoid Arthritis
Brief Title: Natrunix Versus Methotrexate in Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: XBiotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-PT059
Record Dates: First submitted 2022-05-02; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Folic Acid

STUDY DESIGN:
Intervention Model Description: Arm 1: Natrunix with MTX placebo (+folate) Arm 2: Natrunix placebo with MTX (+folate)
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Natrunix with MTX placebo (+Folate) (Experimental): Natrunix 400mg, subcutaneous injection with oral MTX placebo (+Folate). This arm will enroll 100 subjects.
  Interventions: Drug: Natrunix with MTX placebo (+folate)
- Natrunix Placebo with MTX(+Folate) (Active Comparator): Natrunix Placebo, subcutaneous injection with oral MTX(+Folate). This arm will enroll 50 subjects.
  Interventions: Drug: Natrunix placebo with MTX (+folate)

INTERVENTIONS:
Drug: Natrunix with MTX placebo (+folate) — True Human IgG4 monoclonal antibody that neutralizes Interleukin-1α
  Arms: Natrunix with MTX placebo (+Folate)
Drug: Natrunix placebo with MTX (+folate) — Natrunix placebo with MTX (+folate)
  Arms: Natrunix Placebo with MTX(+Folate)

SUMMARY:
Phase II Double-Blinded, Placebo-Controlled Randomized Study Examining the Safety and Efficacy of Natrunix versus MTX (+folate) for the Treatment of Rheumatoid Arthritis

DETAILED DESCRIPTION:
The ACR50 response rate will be determined for Natrunix treatment in comparison with MTX (+folate). There will be a total study population of 150 subjects with 1:1 randomization (75 subjects receiving Natrunix + MTX placebo (+folate) and 75 receiving Natrunix placebo + MTX (+folate)).

Patients will undergo a preliminary assessment for study eligibility. Patients who meet the eligibility criteria will be screened and be required to provide an informed consent to acknowledge understanding and accept enrollment in the clinical study. Subjects enrolled will be randomized in a 1:1 ratio to receive either test article (Natrunix) + MTX placebo OR Natrunix placebo + MTX (+folate). Four weeks are allotted to complete all screening procedures. During the screening period, certain treatments will be washed out (discontinued), as applicable, according to eligibility requirements.

Clinical assessments and collection of blood samples for Natrunix pK determination or other analysis will be performed at specified clinic visits. Natrunix + MTX placebo (+folate) OR Natrunix placebo + MTX (+folate) will be administered weekly for 12 weeks. After 13 weeks, the study will conclude. All data must be entered into the database in a timely manner, including data from the last visit.

Patients will receive the following treatments every week: 400 mg Natrunix or Natrunix placebo injected subcutaneously once a week, followed by MTX placebo or MTX taken orally once a week respectively and a minimum of 1 mg folic acid taken orally every day or 5 mg of folinic acid taken orally once a week.

A patient should start on a reduced dose of 7.5 mg of MTX or MTX placebo at visit 1. On day 5 (5 days after the first dose), the patient laboratory findings are checked and if there are no clinically significant findings, the dose of MTX or MTX placebo may be increased up to 15 mg once weekly and maintained throughout the study. The dose of MTX may range from 7.5-15 mg once weekly based on discretion of the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing comply with MTX regimen (+folate) and have no prior MTX (+folate) intolerance.
* Subject has no prior history of MTX (+folate) failure for the treatment of RA.
* Diagnosis of RA for greater than or equal to 3 months.
* Meets the following minimum disease activity criteria at screening and baseline: ≥6 swollen joints (based on DAS28) and ≥6 tender joints (based on DAS28) and DAS-ESR > 3.2.
* Normal CBC, hepatic and bone marrow function according to the site's institutional guidelines.
* Male or female, at least 18 years, willing to provide informed consent; able to attend all clinic visits and comply with study-related procedures; and able to understand and complete study-related questionnaires.

Exclusion Criteria:

* History of treatment with Natrunix for any reason.
* Uncontrolled intercurrent illness (e.g., ongoing infection, psychiatric illness/social situations that would limit compliance with study requirements).
* Subject has a prior history of MTX (+folate) failure for the treatment of RA.
* Subjects received MTX (+folate) for any reason for the previous 6 weeks prior to randomization.
* Patients must not have received any biological therapy within 8 weeks prior to randomization.
* No treatment with protein tyrosine kinase (PTK) inhibitors within 4 weeks of randomization.
* Investigational therapy administered within a time interval less than at least 5 half-lives of the investigational agent, whichever was longer, prior to the first scheduled day of dosing in this study.
* Pregnant or breastfeeding subjects.
* Patients with alcoholism or other substance abuse.
* Uncontrolled heart disease, including NYHA Class III or IV congestive heart failure, ventricular arrhythmias, uncontrolled blood pressure (defined as ≥ 160/100 mm Hg), or unstable angina.
* Any other concomitant disease, disorder, or condition that could interfere with patient's safety, ability to participate, or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
ACR 50 response rate at 12 weeks. | At 12 weeks from baseline
  The ACR is a measure used in clinical practice and clinical trial to assess medication efficacy in patients with RA, by notating improvements in swelling and tenderness in designated joints, as well as improvements in at least 3 out of 5 other categories. The other categories assessed are patient global assessment of disease activity, physician global assessment of disease activity, patient reported pain scale, disability/functionality questionnaire response, and acute phase reactant levels (CRP and ESR).

SECONDARY OUTCOMES:
ACR 20 response rate at 12 weeks. | At 12 weeks from baseline
Mean change in NRS-pain at 12 weeks. | At 12 weeks from baseline
  Numerical rating scale (NRS) is a validated measure used to assess chronic and acute pain using a 10 point rating scale. The rating for no pain is "0" and "worst possible pain" is 10.